CLINICAL TRIAL: NCT06377501
Title: Feasibility of a Whole-Food, Plant-Based Dietary Intervention for Patients With Low-Risk Chronic Lymphocytic Leukemia
Brief Title: Feasibility of a Whole-Food, Plant-Based Diet for Patients With Low-Risk Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Ariel Portera, Assistant Professor Family Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 804687
Record Dates: First submitted 2023-04-05; First posted 2024-04-22 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Chronic Lymphocytic Leukemia Stage A(0)
Keywords: whole-food plant-based diet; CLL
MeSH Terms: interventions — Diet, Plant-Based

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Subjects will be instructed to adopt a whole-food, plant-based diet for 8 weeks. They will attend weekly group cooking classes led by a RD and receive weekly health coaching sessions.
  Interventions: Other: Whole-food, plant-based diet

INTERVENTIONS:
Other: Whole-food, plant-based diet — Subjects will be instructed to adopt a whole-food, plant-based diet for 8 weeks. They will attend weekly group cooking classes led by a RD and receive weekly health coaching sessions.

SUMMARY:
This study will evaluate the feasibility of an 8-week vegan whole-food, plant-based dietary intervention in subjects with low risk CLL who are undergoing observation. Over the course of 8 weeks, participants will attend weekly group cooking classes via Zoom lead by a RD. Participants will also attend weekly individual meetings with a health coaches to assist with adherence to the dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a diagnosis of low-risk CLL according to the modified Rai staging criteria for a minimum of 12 months and are currently undergoing observation.
* Access to a computer or tablet and Zoom.

Exclusion Criteria:

* Have active disease and are currently receiving pharmacologic treatment for CLL
* Have previously received treatment for CLL
* Are currently following a vegan or vegetarian diet
* A previous or current diagnosis of disordered eating including anorexia, bulimia, binge eating disorder or avoidant/restrictive food intake disorder.
* A diagnosis of Type 1 diabetes
* A diagnosis of Insulin dependent type 2 diabetes
* Currently pregnant or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Adherence to the Dietary Intervention | Up to 24 weeks
  Adherence to the dietary intervention will be calculated using a dietary index developed specifically for this diet. Dietary adherence scores will be calculated using a pre- and post-intervention food frequency questionnaire, as well as 3-day food diaries obtained throughout the intervention.
Satisfaction with the Dietary Intervention | 8 weeks
  Subject satisfaction will be assessed post-intervention using an acceptability, appropriateness and feasibility questionnaire. The questionnaire does not use a scoring system, rather statements will be provided and participants will provide an answer ranging from "completely disagree" to "completely agree."
Cooking Class Adherence | 8 weeks
  Cooking class attendance will also be used as a measure of adherence.
Recruitment | Through study completion, an average of 1 year
  Recruitment rate will be assessed by examining the number of potentially eligible participants, number contacted, consent rates, number completing the intervention.
Retention | 8 weeks
  Retention will be calculated using the number of participants who enroll in the study and the number of participants who complete the 8 week intervention.

SECONDARY OUTCOMES:
White blood cell count | Change from baseline at 4 weeks and 8 weeks.
  Will be measured using standard methods.
Absolute lymphocyte count | Change from baseline at 4 weeks and 8 weeks.
  Will be measured using standard methods.
Anthropometric Measures (height, weight, body mass index) | Change from baseline at 4 weeks and 8 weeks.
  Will be measured using standard methods. Weight and height will be combined to report BMI in kg/m^2.
Anthropometric Measures (waist circumference) | Change from baseline at 4 weeks and 8 weeks.
  Will be measured using standard methods. Weight and height will be combined to report BMI in kg/m^2.
Biomarkers of cardiometabolic health (complete metabolic panel) | Change from baseline at 4 weeks and 8 weeks.
  Will be measured using standard methods.
Biomarkers of cardiometabolic health (hemoglobin A1c) | Change from baseline at 4 weeks and 8 weeks.
  Will be measured using standard methods.
Biomarkers of cardiometabolic health (cholesterol and triglycerides) | Change from baseline at 4 weeks and 8 weeks.
  Will be measured using standard methods.
Concentration of vitamin B12 | Change from baseline at 4 and 8 weeks.
  Will be measured using standard methods.
Concentration of vitamin B9 | Change from baseline at 4 and 8 weeks.
  Will be measured using standard methods.
Concentration of iron | Change from baseline at 4 and 8 weeks.
  Will be measured using standard methods.
Concentration of ferritin | Change from baseline at 4 and 8 weeks.
  Will be measured using standard methods.
Blood pressure | Change from baseline at 4 weeks and 8 weeks.
  Will be measured using standard methods, both systolic and diastolic blood pressure will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Portera, DO, Principal Investigator — UC San Diego
Locations (1):
- UC San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT06377501/ICF_000.pdf